CLINICAL TRIAL: NCT03911440
Title: Diagnosis and Treatment of Mycoplasma Pneumoniae and Vaccine Development
Brief Title: Treatment and Vaccine Development of Mycoplasma Pneumoniae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201712045MINA
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Atypical Pneumonia
Keywords: Mycoplasma pneumoniae, Macrolide-resistance, Children
MeSH Terms: conditions — Pneumonia, Mycoplasma | interventions — Doxycycline; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azithromycin (Active Comparator): Azithromycin (10mg/kg/day) is given to children with mycoplasma pneumonia for 3 days.
  Interventions: Drug: Azithromycin
- Doxycycline (Experimental): Doxycycline (2-4mg/kg/day) is given to children with mycoplasma pneumonia for 5-10 days.
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — Oral doxycycline is given with a dosage of 2-4 mg/kg/day divided into twice a day for 5-10 days.
  Arms: Doxycycline
Drug: Azithromycin — Azithromycin is given with a dosage of 10 mg/kg/day once a day for 3 days.
  Arms: Azithromycin

SUMMARY:
A randomized clinical trial comparing treatment effectiveness of azithromycin and doxycycline for pediatric Mycoplasma pneumonia.

DETAILED DESCRIPTION:
Mycoplasma pneumoniae accounts for 10-30% of community-acquired pneumonia (CAP) in children. Proportionally, M. pneumoniae has become the most important pathogen for childhood pneumonia after the widespread use of Streptococcus pneumoniae vaccines. M. pneumoniae is routinely treated with antibiotics, and the macrolides antibiotics are the drug of choice for M. pneumonia infection. However, macrolide-resistance rates have increased to 20 and 100% in Asia. In previous studies, the most common mutation point, A2063G, was detected from 23% of local strains in Taiwan. The evolution and spreading of Mycoplasma in Taiwan and different countries are unknown. While the macrolide-resistance is increasing, the optimal therapy remains unclear. Both tetracyclines and fluoroquinolones showed promises in treating macrolide-resistant M. pneumoniae in adults. However, their use in children is not recommended due to safety concerns. Recently, evidence are accumulating that doxycycline, unlike other tetracyclines, does not cause staining of teeth. In the current study, the investigators are going to carry out a randomized control trial to compare the efficacy and safety of doxycycline against macrolide-resistant M. pneumoniae.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-18 years, admitted due to lower respiratory tract infections. Mycoplamsa pneumonia is diagnosed.
* The diagnosis is made within 72 hours after fever onset.
* The patient and his/her guardians are willing to participate the study and able to follow the instruction.

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Defervescence | Up to 10 days
  The timing (days) when fever subsides after treatment

SECONDARY OUTCOMES:
Hospital stay | Up to 2 weeks
  The length of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No